CLINICAL TRIAL: NCT01251731
Title: A Randomized, Double-Blind, Placebo-Controlled, 3-Way Crossover Study to Evaluate the Single-Dose Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of 10, 40, and 80 mg E5501 Followed by a Selected Dose for Multiple Dosing Administered to Healthy Japanese, Chinese, and Caucasian Subjects
Brief Title: Single and Multiple Dose Asian Bridging Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E5501-A001-006
Record Dates: First submitted 2010-11-30; First posted 2010-12-02 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — avatrombopag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Treatment Group 1 (Experimental)
  Interventions: Drug: E5501
- Treatment Group 2 (Experimental)
  Interventions: Drug: E5501
- Treatment Group 3 (Experimental)
  Interventions: Drug: E5501
- Treatment Group 4 (Experimental)
  Interventions: Drug: E5501

INTERVENTIONS:
Drug: E5501 — Treatment Group 1: 10mg E5501 as a single dose in Treatment Period 1, followed by a single dose of 40mg E5501 in Treatment Period 2, followed by a single dose of 80mg E5501 in Treatment Period 3, followed by a selected dose for the Multiple Dose reatment Period.
  Arms: Treatment Group 1
Drug: E5501 — Treatment Group 2: 40 mg E5501 as a single dose in Treatment Period 1, followed by a single dose of 80mg E5501 in Treatment Period 2, followed by a single dose of 10mg E5501 in Treatment Period 3, followed by a selected dose for the Multiple Dose Treatment Period.
  Arms: Treatment Group 2
Drug: E5501 — Treatment Group 3: 80mg E5501 as a single dose in Treatment Period 1, followed by a single dose of 10mg E5501 in Treatment Period 2, followed by a single dose of 40mg E5501 in Treatment Period 3, followed by a selected dose for the Multiple Dose Treatment Period.
  Arms: Treatment Group 3
Drug: E5501 — Treatment Group 4: A single dose of matching placebo in each of the three Single Dose Treatment Periods and in the Multiple Dose Treatment Period
  Arms: Treatment Group 4

SUMMARY:
The purpose of this study is to evaluate the single-dose (SD) pharmacokinetics (PK), pharmacodynamics (PD), safety and tolerability of 10, 40, and 80 mg E5501 followed by a selected dose for multiple dosing (MD) in healthy Japanese, Chinese, and Caucasian subjects.

DETAILED DESCRIPTION:
This study will evaluate the single-dose (SD) pharmacokinetics (PK), pharmacodynamics (PD), safety, and tolerability of oral doses of 10, 40, and 80 mg E5501 administered to 36 healthy male and female Japanese, Chinese, and Caucasian subjects. For the SD Treatment Period, 12 subjects from each ethnic group will be randomized to receive single doses of 10, 40, or 80 mg E5501 or matching placebo each treatment period. Each subject will be allocated to a treatment sequence to be dosed with either placebo for the three periods or dosed with each of the three different doses in the three periods. For the Multiple-Dose (MD) Treatment Period the 12 subjects in each ethnic group will be further randomized as active (dose level to be determined from the SD Treatment Period or placebo in a 3:1 ratio.

ELIGIBILITY:
Key Inclusion Criteria:

* Normal healthy adult males and females (age 20-45 years)
* Body Mass Index greater than or equal to 18 and less than or equal to 29 at the time of screening
* Japanese and Chinese subjects must be born in their respective countries of origin and have parents and grandparents of Japanese or Chinese descent, respectively
* Japanese subjects must have lived outside of Japan for no more than 5 years; Chinese subjects must have lived outside of China for no more than 10 years
* In addition to mainland China, Chinese subjects may be from Taiwan, Hong Kong, or Mongolia
* Japanese and Chinese subjects must not have significantly changes their lifestyle with regard to diet; i.e., their diet must not have significantly changed since leaving China or Japan
* Platelet count between 150,000 and 300,000/mm3

Key Exclusion Criteria:

* Evidence of clinically significant cardiovascular, hepatic, gastrointestinal, renal, respiratory, endocrine, hematologic, neurologic, or psychiatric disease or abnormalities or a known history of any gastrointestinal surgery that could impact the PK of the study drug
* Evidence of organ dysfunction or any clinically significant deviation from normal in their medical history, e.g., history of splenectomy
* History of venous or arterial thrombotic disease or other hypercoagulable state
* Hemoglobin level less than 12.0 g/dL

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2010-07; Primary Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
• To compare the single-dose pharmacokinetics (PK), as measured by AUCinf of three doses of E5501 (10, 40, and 80 mg) in healthy Japanese and Chinese subjects relative to healthy Caucasian subjects | up to 96 hours post-dose
• To compare the multiple-dose steady-state PK, as measured by AUCss, of E5501 in healthy Japanese and Chinese subjects relative to Caucasian subjects | up to 96 hours after dosing on Day 7 or up to 240 hours after the first drug dosing
• To compare the multiple-dose pharmacodynamic (PD) response as measured by platelet counts for E5501 in healthy Japanese and Chinese subjects relative to Caucasian subjects | through Day 21 for each SD Treatment Period and through Day 30 for the MD Treatment Period
• To compare the single-dose pharmacokinetics (PK), as measured by Cmax of three doses of E5501 (10, 40, and 80 mg) in healthy Japanese and Chinese subjects relative to healthy Caucasian subjects | up to 96 hours post-dose

SECONDARY OUTCOMES:
To evaluate single-dose linearity of 10, 40 and 80mg E5501 in healthy Japanese, Chinese, and Caucasian subjects | from Day 1 SD Treatment Period 1 through Day 30 MD Treatment Period 4
To characterize PK/PD relationships between E5501 exposure and platelet count response in healthy Japanese, Chinese, and Caucasian subjects | from Day 1 SD Treatment Period 1through Day 30 MD Treatment Period 4

CONTACTS AND LOCATIONS:
Overall Officials: Franklin Johnson, Study Director — Eisai Inc.
Locations (1):
- Parexel International, Early Phase Clinical Unit, Los Angeles, California, United States